CLINICAL TRIAL: NCT03857009
Title: Why Does my Shoulder Hurt? Identifying Factors Associated With the Presence of Pain in Individuals With Full-thickness Rotator Cuff Tears
Brief Title: Why Does my Shoulder Hurt? Understanding the Presence of Pain in Individuals With Full-thickness Rotator Cuff Tears
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Associate Professor, Faculty of Medicine, Laval University
Other Study IDs: ShoulderPain2018
Record Dates: First submitted 2018-08-09; First posted 2019-02-27 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Full-thickness Rotator Cuff Tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA (saliva) samples will be collected at the baseline evaluation only. The samples will be analyzed for pain modulatory genes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic: No intervention.
- Asymptomatic: No intervention.

SUMMARY:
Full-thickness rotator cuff tears (FTRCT), defined as "through-and-through" tears of one of the shoulder tendons, affect up to 32% of the population (mostly individuals older than 50 years) and are one of the most painful and debilitating shoulder diagnoses. One of the primary challenges for clinical decision-making is the poor association between the presence of FTRCT (detected by medical imaging) and pain, as studies have shown that 2/3 of people with FTRCT are asymptomatic. This challenges the notion that FTRCT causes pain, and highlights the fact that symptoms may be explained by other variables. A better understanding of the factors leading to the development of pain in people with FTRCT would optimize clinical care (including prevention).

The objective of this study is to identify variables associated with pain in people with FTRCT by 1) comparing people with FTRCT with (Symptomatic Group; n=40) and without pain (Asymptomatic Group; n=40); 2) comparing people who initially have pain-free FTRCT (Asymptomatic Group) who develop pain over a 2-year period to those who do not develop pain; and 3) comparing people who initially have painful FTRCT (Symptomatic Group) who become pain-free over a 2-year period to those who remain symptomatic. All participants will undergo an ultrasound examination to confirm the presence of FTRCT, and information on a number of variables (sociodemographic, anatomical, genetic, psychosocial, pain sensitivity, neuromuscular, biomechanical) will be collected. All participants will then be followed for 2 years before being revaluated for pain. Variables will be analysed to determine those associated with pain. As it is crucial to improve our understanding of the mechanisms leading to pain, this project has the potential to impact the musculoskeletal health of Canadians. By considering multiple variables associated with FTRCT, its results could lead to the development of tangible solutions to optimize prevention and recovery.

DETAILED DESCRIPTION:
Background: Symptomatic full-thickness rotator cuff tears (FTRCT) affect up to 32% of the population and represent one of the more painful and debilitating shoulder diagnoses. The prevailing model for care pathway decisions is heavily influenced by medical imaging. Yet, the association between FTRCT observed on medical imaging and the presence of pain is poor, as two thirds of FTRCT are asymptomatic. This poses a great challenge to clinical decision-making and questions the belief that FTRCT causes pain. As other factors may explain the presence of pain, a better understanding of this phenomenon needs to be sought.

Objective/hypothesis: The primary objective is to identify variables associated with the presence of pain in individuals with FTRCT. The hypothesis is that given its complex aetiology, no single outcome will be highly associated with pain, rather it will be important to consider several outcomes and their interactions. Secondary objectives include: to explore if a) baseline variables or b) a change in these variables following baseline can predict the development of pain in individuals who initially have asymptomatic FTRCT, and to study if a) baseline variables or b) a change in these variables following baseline can predict the resolution of pain in individuals who initially have symptomatic FTRCT.

Methods: 40 adults with a FTRCT and shoulder pain (Symptomatic Group), and 40 adults with a FTRCT without shoulder pain (Asymptomatic Group) will be included. They will demonstrate a FTRCT on US examinations performed by a radiologist. Included participants will take part in a baseline evaluation during which sociodemographic, anatomical, genetic, psychosocial, pain sensitivity, neuromuscular and biomechanical variables will be assessed. The primary objective (cross-sectional design) will be achieved by determining if differences between groups are based on a sole or on several independent variables, and their relative impact on pain (recursive partitioning, principal component analysis, MANOVA).

The secondary objectives (prospective design) will be achieved by following all participants for 2 years. Every 3 months, the participants will complete a web-based questionnaire asking if they have had shoulder pain. Participants in the Asymptomatic Group who develop pain and participants in the Symptomatic Group who become pain-free will be asked to participate in a follow-up evaluation within a week. Participants who remain pain-free in the Asymptomatic Group and with pain in the Symptomatic Group during the follow-up period will also be asked to participate in a follow-up evaluation at the end of the 2 years (same follow-up evaluation for all participants, similar to baseline evaluations). Logistic regressions will be used to identify the variables associated with pain development and with pain resolution.

Relevance: Before implementing new intervention strategies, a better understanding of factors associated with the presence of pain is needed. By looking at different variables that could explain pain, this project will improve our understanding of FTRCT and fill important knowledge gaps.

ELIGIBILITY:
Inclusion Criteria (all participants):

* Presence of a full-thickness rotator cuff tear (on ultrasound examination performed by a radiologist)
* 50 to 80 years of age
* Degenerative tear (no significant trauma)

Inclusion Criteria for the Symptomatic group:

* unilateral or bilateral shoulder pain (at least 2/10 on a visual analog scale [VAS] evaluating usual shoulder pain)
* positive response to: 'In the past 4 weeks, have you had pain in your shoulder' and 'If yes, was this pain bad enough to limit your usual activities or change your daily routine for more than 1 day?'

Inclusion Criteria for the Asymptomatic group:

* report no current shoulder pain (0/10 on a VAS evaluating usual shoulder pain)
* negative response to: 'In the past 4 weeks, have you had pain in your shoulder'
* do not report any past significant shoulder pain (any pain greater than or equal to 2/10 that lasted longer than 4 weeks, required the use of medications or prompted a physician visit)

Exclusion Criteria:

1. unable to understand French or English;
2. history of upper limb fracture;
3. previous shoulder surgery;
4. cervicobrachialgia or shoulder pain reproduced by neck movement;
5. shoulder capsulitis (restriction of at least 30% in 2 or more directions);
6. rheumatoid, inflammatory or neurological diseases;
7. corticosteroid injection in the previous 6 weeks;
8. cognitive problems interfering with evaluations (Mini-Mental State Examination ≥ 24)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 50 to 80 years presenting with symptomatic or asymptomatic full-thickness rotator cuff tears.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in usual shoulder pain from baseline: Visual analog scale (VAS) | From baseline to the follow-up evaluation (end of the 2-year period) (Objective 2 and 3)
  Participants will be asked to rate the intensity of their pain on a VAS from 0 to 10, where "0" represents no pain and "10" represents "worst pain imaginable", in the last week, month and 3 months. Highest possible score (worst outcome): 30. Lowest possible score (best outcome): 0. Method to compute total score: sum of each score.
usual shoulder pain from baseline: Visual analog scale (VAS) | Baseline score (Objective 1)
  Participants will be asked to rate the intensity of their pain on a VAS from 0 to 10,

SECONDARY OUTCOMES:
Change from baseline with regard to: Sociodemographic and occupational factors | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  General sociodemographic questionnaire including sex; gender; date of birth; age; height; weight; hand dominance; racial, ethnic or cultural origin; civil status; education level; occupation; employment status; overhead sports activities (currently or previously); household income; smoking habits
Sociodemographic and occupational factors | Baseline characteristics (Objective 1)
  General sociodemographic questionnaire including sex; gender; date of birth; age; height; weight; hand dominance; racial, ethnic or cultural origin; civil status; education level; occupation; employment status; overhead sports activities (currently or previously); household income; smoking habits
Change in disability and functional limitations of the upper extremity from baseline: QuickDASH | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Questionnaire comprising 11 questions evaluating disability and functional limitations of the upper extremity on a scale from 1 to 5, where 1 denotes full capacity and 5 denotes incapacity
Disability and functional limitations of the upper extremity QuickDASH | Baseline score (Objective 1)
  Questionnaire comprising 11 questions evaluating disability and functional limitations of the upper extremity on a scale from 1 to 5, where 1 denotes full capacity and 5 denotes incapacity
Change in comorbidities from baseline: Self-Administered Comorbidity Questionnaire | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Questionnaire determining the presence or absence of 13 health problems, whether or not the person is treated for each problem, and whether or not the problem interferes with / limits their activities
Comorbidities: Self-Administered Comorbidity Questionnaire | Baseline score (Objective 1)
  Questionnaire determining the presence or absence of 13 health problems, whether or not the person is treated for each problem, and whether or not the problem interferes with / limits their activities
Change in sleep disturbance from baseline: PROMIS Sleep Disturbance Questionnaire | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Qualitative questionnaire on a 5-point Likert scale, where higher scores indicate greater sleep quality
Sleep disturbance: PROMIS Sleep Disturbance Questionnaire | Baseline score (Objective 1)
  Qualitative questionnaire on a 5-point Likert scale, where higher scores indicate greater sleep quality
Change in prevalence and frequency of symptoms from baseline: Nordic Musculoskeletal Questionnaire | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Questionnaire evaluating the prevalence of pain (dichotomous scale, "yes" or "no") in all regions of the body (in the last week, last 3 months and last 12 months), and the frequency of pain/symptoms in each region of the body (scale from 0 to 3, where higher scores indicate higher frequency of symptoms)
Prevalence and frequency of symptoms from baseline: Nordic Musculoskeletal Questionnaire | Baseline score (Objective 1)
  Questionnaire evaluating the prevalence of pain (dichotomous scale, "yes" or "no") in all regions of the body (in the last week, last 3 months and last 12 months), and the frequency of pain/symptoms in each region of the body (scale from 0 to 3, where higher scores indicate higher frequency of symptoms)
Change in anxiety from baseline: State-Trait Anxiety Inventory | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  6 items each scored on a 4-point scale, higher scores denote greater anxiety
Anxiety from baseline: State-Trait Anxiety Inventory | Baseline score (Objective 1)
  6 items each scored on a 4-point scale, higher scores denote greater anxiety
Change in depressive symptoms from baseline: Patient Health Questionnaire | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  9-item questionnaire evaluating depressive symptoms, on a 4-point scale where higher scores denote higher frequency of depressive symptoms
Depressive symptoms from baseline: Patient Health Questionnaire | Baseline score (Objective 1)
  9-item questionnaire evaluating depressive symptoms, on a 4-point scale where higher scores denote higher frequency of depressive symptoms
Change in perceived stress from baseline: Perceived Stress Scale 4 | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  4-item questionnaire, scored on a 5-point scale from 0 ("never") to 4 ("very often"). Higher scores are correlated to more stress.
Perceived stress from baseline: Perceived Stress Scale 4 | Baseline score (Objective 1)
  4-item questionnaire, scored on a 5-point scale from 0 ("never") to 4 ("very often"). Higher scores are correlated to more stress.
Change in upper extremity work demands from baseline: Revised Upper Extremity Work Demands Scale (currently and previously) | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  6-item scale scored from 1 ("rarely / never") to 4 ("almost always"), higher scores indicate greater physical work demands on the upper extremity.
Upper extremity work demands from baseline: Revised Upper Extremity Work Demands Scale (currently and previously) | Baseline score (Objective 1)
  6-item scale scored from 1 ("rarely / never") to 4 ("almost always"), higher scores indicate greater physical work demands on the upper extremity.
Change in pain catastrophising from baseline: Pain Catastrophising Scale | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  13-item questionnaire, 5-point scale, greater scores indicate more pain catastrophizing.
Pain catastrophising from baseline: Pain Catastrophising Scale | Baseline score (Objective 1)
  13-item questionnaire, 5-point scale, greater scores indicate more pain catastrophizing.
Change in Structural tissue damage of the shoulder from baseline (ultrasound evaluation performed by a radiologist) | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Full thickness rotator cuff tears will be classified by size defined as small (<10 mm), medium (10 to 30 mm) or large (>30 mm)
Structural tissue damage of the shoulder from baseline (ultrasound evaluation performed by a radiologist) | Baseline observations (Objective 1)
  Full thickness rotator cuff tears will be classified by size defined as small (<10 mm), medium (10 to 30 mm) or large (>30 mm)
Change in Acromiohumeral distance from baseline | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Ultrasound (US scanner) will be used to measure the acromiohumeral distance of the affected shoulder at 0 degrees and 60 degrees of shoulder abduction
Acromiohumeral distance from baseline | Baseline distance (Objective 1)
  Ultrasound (US scanner) will be used to measure the acromiohumeral distance of the affected shoulder at 0 degrees and 60 degrees of shoulder abduction
Change in Radiographical evaluation of the shoulder from baseline | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Presence or absence of calcific tendonitis and/or osteophytes at the glenohumeral and acromioclavicular joints
Radiographical evaluation of the shoulder from baseline | Baseline observation (Objective 1)
  Presence or absence of calcific tendonitis and/or osteophytes at the glenohumeral and acromioclavicular joints
Change in pain sensitivity from baseline: Pressure Pain Threshold (PPT) | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  PPT will be assessed bilaterally at the middle deltoid and tibialis anterior muscles using a mechanical pressure algometer at an applied rate of 1 kg/s. The amount of pressure at which pain is perceived (in Newtons) will be recorded (mean of 3 trials). Higher scores denote less pain sensitivity.
Pain sensitivity from baseline: Pressure Pain Threshold (PPT) | Baseline score (Objective 1)
  PPT will be assessed bilaterally at the middle deltoid and tibialis anterior muscles using a mechanical pressure algometer at an applied rate of 1 kg/s. The amount of pressure at which pain is perceived (in Newtons) will be recorded (mean of 3 trials). Higher scores denote less pain sensitivity.
Change in Range of Motion (ROM) of the affected shoulder from baseline | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Shoulder ROM in flexion, lateral rotation at 0° abduction, and lateral and medial rotation at 90° abduction will be measured using a goniometer (flexion) and an inclinometer (other measures). Values will be compared to normative data according to age.
Range of Motion (ROM) of the affected shoulder from baseline | Baseline ROM (Objective 1)
  Shoulder ROM in flexion, lateral rotation at 0° abduction, and lateral and medial rotation at 90° abduction will be measured using a goniometer (flexion) and an inclinometer (other measures). Values will be compared to normative data according to age.
Change in Bilateral grip strength with handheld dynamometer from baseline | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Measured in pounds.
Bilateral grip strength with handheld dynamometer from baseline | Baseline score (Objective 1)
  Measured in pounds.
Change in Isometric shoulder strength from baseline, with manual dynamometer | BFrom baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Isometric shoulder strength in abduction and in lateral rotation at 0° abduction will be measured in Newtons with a manual dynamometer (MedUp), and normalized by lever arm, measured in meters using a measuring tape.
Isometric shoulder strength from baseline, with manual dynamometer | Baseline score (Objective 1)
  Isometric shoulder strength in abduction and in lateral rotation at 0° abduction will be measured in Newtons with a manual dynamometer (MedUp), and normalized by lever arm, measured in meters using a measuring tape.
Change in scapular dyskinesis from baseline: Scapula Dyskinesis Test | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Bilateral scapular dyskinesis measured on a 3-point scale: normal (0 points), subtle (1 point), obvious (2 points). Higher scores indicate greater dyskinesis.
Scapular dyskinesis from baseline: Scapula Dyskinesis Test | Baseline score (Objective 1)
  Bilateral scapular dyskinesis measured on a 3-point scale: normal (0 points), subtle (1 point), obvious (2 points). Higher scores indicate greater dyskinesis.
Change from baseline in Shoulder proprioception (arm position matching), coordination and functional dominance with the KINARM exoskeleton (BKIN Technologies) | From baseline to the follow-up evaluation (end of the 2-year period)(Objective 2 and 3)
  Three KINARM standard tasks will be used to evaluate bilateral upper extremity neuromuscular control. Units of measurement: error in cm and task score (arm position matching task), and task score for the coordination and functional dominance tasks. Task scores are calculated by KINARM software according to variables such as precision and speed.
Shoulder proprioception (arm position matching), coordination and functional dominance with the KINARM exoskeleton (BKIN Technologies) | Baseline score (Objective 1)
  Three KINARM standard tasks will be used to evaluate bilateral upper extremity neuromuscular control. Units of measurement: error in cm and task score (arm position matching task), and task score for the coordination and functional dominance tasks. Task scores are calculated by KINARM software according to variables such as precision and speed.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PT, PhD, Principal Investigator — Laval University
Locations (1):
- Center for Interdisciplinary Research in Rehabilitation and Social Integration (CIRRIS), Québec, Quebec, Canada